CLINICAL TRIAL: NCT04940962
Title: Translational Study Using Human Abdominal Adipose Tissue Biopsies to Investigate the Role of Cannabinoid Receptor 1 (CB1) in Controlling Endocannabinoid and Adipokine Secretion
Acronym: ENDOCATA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VERGES 2020
Record Dates: First submitted 2021-05-10; First posted 2021-06-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Diabete Type 2; Abdominal Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Non-diabetic obese (Experimental)
  Interventions: Procedure: Sampling of adipose tissue
- Diabetic obese (Experimental)
  Interventions: Procedure: Sampling of adipose tissue
- Witnesses (Active Comparator)
  Interventions: Procedure: Sampling of adipose tissue

INTERVENTIONS:
Procedure: Sampling of adipose tissue — Removal of less than 1 cm3 of adipose tissue during visceral surgery

SUMMARY:
Abdominal obesity and type 2 diabetes are associated with the hyperactivation of the endocannabinoid system. Several animal and human studies indicate that circulating endocannabinoid (EC) levels are correlated with body fat. Thus, adipose tissue, which possesses the enzymatic machinery for the synthesis of ECs, could be the main producer of plasma ECs.

Today, it is clearly established that stimulation of the endocannabinoid system, via activation of cannabinoid receptor 1 (CB1s) located in the brain, leads to increased food intake and weight gain. Moreover, peripheral CB1s present in organs such as the liver, muscles and adipose tissue are involved in the establishment of metabolic deregulations linked to obesity (steatosis, insulin resistance, dyslipidemia).

Thus, ECs produced by adipose tissue could play a key role in the regulation of carbohydrate-lipid homeostasis through their autocrine or paracrine actions by activating central and peripheral CB1s. Therefore, the objective of this study is to:

1. clarify whether obesity, associated or not with diabetes, leads to an overproduction of ECs (specifying which ones) by visceral or subcutaneous adipose tissue
2. to determine whether blocking CB1s with new peripherally acting antagonists can lead to a reduction in the production of ECs by adipose tissue.

This study will also provide an opportunity to evaluate the production of adipokines and cytokines involved in the control of energy homeostasis under the different experimental conditions.

ELIGIBILITY:
Inclusion Criteria:

* Controls:
* men or post-menopausal women aged between 18 and 80
* gave oral consent
* to undergo visceral surgery

Non-diabetic obese subjects:

* men or post-menopausal women aged between 18 and 80
* BMI > 30
* gave oral consent
* to undergo visceral surgery

Obese diabetic subjects:

* men or post-menopausal women aged between 18 and 80
* type 2 diabetic not treated with Insulin or GLP-1 agonist
* BMI > 30
* gave oral consent
* to undergo visceral surgery

Exclusion Criteria:

* Controls:
* Person not covered by national health insurance.
* BMI > 30
* diabetes
* chronic inflammatory disease
* cancer undergoing chemotherapy or chemotherapy less than a year old
* digestive cancer with recent weight loss (≥10%) and/or malnutrition
* known metastatic cancer
* cancer undergoing long-term hormonal treatment
* protected adult

Non-diabetic obese subjects:

* Person not covered by national health insurance
* diabetes
* chronic inflammatory disease
* cancer undergoing chemotherapy or chemotherapy less than a year old
* digestive cancer with recent weight loss (≥10%) and/or malnutrition
* known metastatic cancer
* cancer undergoing long-term hormonal treatment
* protected adult

Obese diabetic subjects:

* Person not covered by national health insurance
* chronic inflammatory disease
* cancer undergoing chemotherapy or chemotherapy less than a year old
* digestive cancer with recent weight loss (≥10%) and/or malnutrition
* known metastatic cancer
* cancer undergoing long-term hormonal treatment
* type 1 diabetes
* secondary diabetes
* protected adult

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Kinetics of the appearance of endocannabinoids produced by visceral adipose tissue explants in culture medium estimated by the area under the curve in obese subjects and in controls. | 12 hours
  The assay will be performed using a technique of liquide chromatography coupled to a mass spectrometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No